CLINICAL TRIAL: NCT05661214
Title: The Effect of Using Clinical Decision Support System in Pressure Injury Risk Management Teaching of Nursing Students: A Randomized Controlled Study
Brief Title: The Effect of Using Clinical Decision Support System in Pressure Injury Risk Management Teaching
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ozlem Ariburnu, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NI 21/633
Record Dates: First submitted 2022-12-05; First posted 2022-12-22 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Students, Nursing
Keywords: pressure injury risk management; nursing student; randomized controlled trial
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: This study was designed with Solomon four groups design. There will be control group one, control group two, intervention group one and intervention group two.
Who Masked: Participant, Outcomes Assessor
Masking Description: In this study, whole participants will be masked during the study. After study, researchers will encode the data different names and send to the statistician. Therefore, statistician will not know which group is control or intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group 1 (No Intervention): This group is the control group 1 (one) that will be taught using structured standard teaching content. Before teaching, participants will be applied pre tests. After teaching, they will be applied post tests.
- Intervention Group 1 (Experimental): This group is the intervention group 1 (one) that will be taught using model-based structured teaching content. In this teaching content, researchers will teach pressure injury risk factors; after teaching, participants will plan nursing interventions with Clinical Decision Support System (CDSS) integrated software. Before teaching, participants will be applied pre tests. After teaching, they will be applied post tests.
  Interventions: Other: Teaching
- Control Group 2 (No Intervention): This group is the control group 2 (two) that will be taught using structured standard teaching content. After teaching, they will be applied post tests. This group has no pre-test and will be created to increase internal validity, only.
- Intervention Group 2 (Experimental): This group is the intervention group 2 (two) that will be taught using model-based structured teaching content. In this teaching content, researchers will teach pressure injury risk factors; after teaching, participants will plan nursing interventions with Clinical Decision Support System (CDSS) integrated software. After teaching, they will be applied post tests. This group has no pre-test and will be created to increase internal validity, only.
  Interventions: Other: Teaching

INTERVENTIONS:
Other: Teaching — The intervention in this study is teaching. Researchers, will create a pressure injury teaching content and assess this effectiveness and also, intervention groups will use Clinical Decision Support System (CDSS) as a tool to plan nursing interventions.
  Arms: Intervention Group 1; Intervention Group 2

SUMMARY:
The goal of this randomized controlled study is to compare the changes in cognitive, attitudinal and psychomotor domains for pressure injury between nursing students who take model-based structured pressure injury risk management teaching by examining risk factors and plan nursing interventions through sample cases with Clinical Decision Support System (CDSS) integrated software, and nursing students who plan nursing interventions through sample cases on the software by receiving standard teaching. The hypothesis are:

H1: The knowledge of the students who received the model-based structured pressure injury risk management teaching with the CDSS integrated method is different from the control group who received the standard training.

H1a: The attitudes of the students who received the model-based structured pressure injury risk management instruction with the CDSS integrated method to prevent injuries are different from the control group who received the standard training.

H1b: The nursing interventions planned by the students who received the model-based structured pressure injury risk management education with the CDSS integrated method are different from the control group who received the standard education.

DETAILED DESCRIPTION:
The goal of this randomized controlled study is to compare the changes in cognitive, attitudinal and psychomotor domains for pressure injury between nursing students who take model-based structured pressure injury risk management teaching by examining risk factors and plan nursing interventions through sample cases with Clinical Decision Support System (CDSS) integrated software, and nursing students who plan nursing interventions through sample cases on the software by receiving standard teaching.

Method: This randomized controlled trial was planned with two years of nursing students. The study's eligibility criteria are the nursing student must have completed the Fundamentals of Nursing course and clinical practice of this course. The study consists of preparation and implementation phases. The preparation phase consists of the preparation of the training content and software. Researchers will prepare training content and send them to academicians and clinicians who are experts in their fields. Researchers collaborate with software developers to develop the software. After the researchers listed the students who accepted to participate in the study, Students will be randomly assigned to 2 control and two intervention groups by a third researcher who was not involved in the study. The implementation phase of the research will begin with establishing control and intervention groups.

The researchers will first apply the " Pressure Ulcer Prevention Knowledge Assessment Instrument, "Attitude Towards Pressure Ulcer Prevention Instrument " and test case (the pre-tests) to the control 1 group. After that, they will give formal training to both control groups for four weeks and apply the post-tests in the fifth week. They will prepare the nursing care plan, one of the last tests, by analyzing the case via software. After the training of the control groups, the training of the intervention groups will begin. First of all, the intervention 1 group will apply the "Pressure Ulcer Prevention Knowledge Assessment Instrument," "Attitude Towards Pressure Ulcer Prevention Instrument" and the test case (the pre-tests). Afterward, four-week structured training will be given to intervention groups, and post-tests will be applied in the fifth week. They will prepare the nursing care plan, one of the last tests, by analyzing the case through the software integrated with Clinical Decision Support System.

ELIGIBILITY:
Inclusion Criteria:

* The nursing student must be completed Fundamentals of Nursing course and its clinical practices.

Exclusion Criteria:

* The nursing student cannot be a part of this study, if she/he graduated high school/associate degree about health department and work as a health professional.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-10-02 (Estimated); Primary Completion 2024-01-22 (Estimated); Study Completion 2024-01-22 (Estimated)

PRIMARY OUTCOMES:
Knowledge levels of nursing students about pressure injury | 2.5 months (10 weeks)
  The first data, will be obtained with the valid and reliable instrument before teaching period (pre-test). After applying the instrument, researchers will teach the nursing students for five weeks. After, the teaching process is over, researchers will apply the same instrument (post-test) to obtain the data of knowledge. The aim is to determine the rate of change in the knowledge levels of nursing students before and after the education.
Attitudes of nursing students about pressure injury | 2.5 months (10 weeks)
  The first data, will be obtained with the valid and reliable instrument before teaching period (pre-test). After applying the instrument, researchers will teach the nursing students for five weeks. After, the teaching process is over, researchers will apply the same instrument (post-test) to obtain the data of attitude. The aim is to determine the rate of change about the attitudes of nursing students before and after the education.
Psychomotor development of nursing students about pressure injury | 2.5 months (10 weeks)
  The first data, will be obtained with the case and nursing care plan before teaching period (pre-test). After applying the instrument, researchers will teach the nursing students for five weeks. After, the teaching process is over, researchers will apply the same case and nursing care plan (post-test) to obtain the data of psychomotor development. The aim is to determine the rate of change about the psychomotor development of nursing students before and after the education.

CONTACTS AND LOCATIONS:
Overall Officials: Ozlem Ariburnu, Principal Investigator — Hacettepe University

IPD SHARING:
Plan to Share IPD: Undecided